CLINICAL TRIAL: NCT05351060
Title: Implementing a Novel Splinting Technique Using 3D Models for Patients With Scleroderma and Arthritis: A Pilot Study
Brief Title: Novel Splinting Technique Using 3D Models
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Giovanna Fichera (Other)
Collaborators: Precision Valve Automation (Unknown); St Peters Health Partners (Unknown); Ann Steffens Scleroderma Foundation (Unknown); Russell Sage College (Other)
Responsible Party: Sponsor-Investigator, Giovanna Fichera, Co-Investigator, Russell Sage College
Organization: Russell Sage College (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-1019-1
Record Dates: First submitted 2022-03-26; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Arthritis; Osteoarthritis Hand; Scleroderma, Systemic; Scleroderma, Diffuse; Rheumatoid Arthritis
Keywords: Splints; Occupational Therapy, Hand; Printing, Three-Dimensional; Contracture; Rheumatology; Ulcer; Orthotic Devices; Range of Motion, Articular
MeSH Terms: conditions — Arthritis; Scleroderma, Systemic; Scleroderma, Diffuse; Arthritis, Rheumatoid; Contracture; Ulcer | interventions — Orthotic Devices

STUDY DESIGN:
Intervention Model Description: The study will include up to 10 patients with autoimmune diseases, including either scleroderma, rheumatoid arthritis, or osteoarthritis, which may include the elderly. The study will compare pre and post-evaluation measures for each individual participant through a multiple time series design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D model splinting intervention group (Experimental): The researcher will scan the participant's forearm, wrist, and hand with an iPhone camera through the Comb O&P Scan App. Scans will be completed individually to maintain privacy. The entire Comb O&P platform is HIPAA compliant. The data is de-identified encrypted when it moves from the iPhone app to the computer through the cloud. Precision Valve Automation (PVA) will use the de-identified scans to print the 3D models which are a precise replica of the participant's hand. Once the researcher obtains the 3D models, resting hand splints will be fabricated on the 3D models to provide custom-made hand splint(s) to each participant. The participants will receive the splint(s) to wear during the hours of sleep for six weeks.
  Interventions: Other: Custom Fabricated Splint

INTERVENTIONS:
Other: Custom Fabricated Splint — Participants will wear a customized splint on their affected hand(s)during the hours of sleep for the duration of the study.
  Other Names: Orthotic

SUMMARY:
The purpose of the study is to determine the feasibility of a non-contact custom splint fabrication method for patients with chronic diseases suffering from hypersensitive skin or compromised skin integrity. Custom splinting by occupational therapists involves molding low-temperature thermoplastic material directly on patients' skin; however, skin sensitivity is a contraindication for splint fabrication. The study aims to recruit 10 male or female patients with either a diagnosis of scleroderma (SSc) or arthritis. A scan of the patient's hand and a 3D printer will be used to create a precise model of a patient's hand on which a custom splint will be fabricated. By taking this approach, traditional splinting is substituted by avoiding direct contact with the material on the surface of the patient's upper extremity. This technique creates therapeutic opportunities for underserved patients by expanding splinting options for patients with scleroderma and arthritis, and addressing the challenges associated with managing chronic diseases.

DETAILED DESCRIPTION:
Arthritis is an inflammatory disease that occurs in the joints of the body. Scleroderma is a disease of the autoimmune system in which the body produces excess collagen in the skin and organs. Depending upon a patient's needs, occupational therapists (OTs) make custom hand splints to support individual goals and promote independence. Conventional splinting methods involve molding low-temperature thermoplastic material directly on a patients' skin; however, many chronic diseases including arthritis and scleroderma carry a predisposition for skin sensitivity or compromised skin integrity, leaving these populations with no alternative. The study will recruit 10 male or female patients with either a diagnosis of arthritis or scleroderma for a 14-week study. Researchers will use a scanner and 3D printer to create a model of a patient's hand prior to splinting, which will allow therapists to custom-fit the 105-degree splinting material on the model. Traditional splinting is substituted by avoiding fabricating the splint directly on the patient's hand and providing the opportunity for patients with hypersensitive skin to benefit from a custom-made splint. Implementing this technique creates opportunities by expanding splinting options for patients with chronic diseases. The goals of this study are to evaluate effectiveness, support positive engagement in daily activities, improve patient outcomes, and promote best practice. The research will also establish a foundation for future studies with custom splinting using 3D printed material.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of either scleroderma, osteoarthritis, or rheumatoid arthritis
* Must have the potential to benefit from wearing a resting hand splint as determined by a certified hand therapist
* Over 18 years of age
* Fluent in English

Exclusion Criteria:

* Patients exhibiting any open wounds on their hands or forearms
* Exhibiting impaired decision making and ability to understand splint care and wear instructions as determined by the ability to answer the questions the student researcher asks after the participant has reviewed the splint education handout
* Under 18 years of age
* Unable to secure reliable transport for the duration of the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-05-16 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-08-19 (Estimated)

PRIMARY OUTCOMES:
Change in range of motion of the hand (measured with a goniometer) | During the initial visit (two weeks before the intervention begins) and again during the second clinical visit (the day before the intervention begins)
  The active range of motion of the participant's affected forearm, wrist, and fingers will be assessed with a goniometer. A change in range of motion across two weeks is being assessed (before the intervention begins).
Change in range of motion of the hand (measured with a goniometer) | Every other week throughout the intervention period, a total of three times during the intervention which is six weeks long.
  The active range of motion of the participant's affected forearm, wrist, and fingers will be assessed with a goniometer. A change in range of motion across the six week intervention period will be assessed.

SECONDARY OUTCOMES:
Change of reported comfort level (in hand) measured through a survey | During the initial visit (two weeks before the intervention begins) and again during the second clinical visit (the day before the intervention begins)
  Patients will document their perceived comfort level in their affected hand in a questionnaire twice, across two weeks, before the study intervention begins. The scale is 0-10. 0 being least uncomfortable to 10 being very comfortable. The change in comfort across two weeks is being assessed before the intervention begins.
Change of reported comfort level (in hand) measured through a survey | Daily throughout the six week intervention period
  Patients will report their perceived comfort level in their hand each morning after wearing the splint in an online or hard copy questionnaire. The scale is 0-10. 0 being least uncomfortable to 10 being very comfortable. The change in comfort in the hand across the six week intervention period is being assessed.
Change in hours of sleep measured through a survey | During the initial visit (two weeks before the intervention begins) and during the second clinical visit (the day before the intervention begins)
  Participants will log their hours of sleep and hours they wear their splint each night to determine if they are able to sleep longer when wearing the splint compared to before they wore the splint. This data will be tracked to ensure the intervention is not decreasing hours of sleep significantly. The change in hours of sleep across two weeks (before the intervention begins) will be assessed.
Change in hours of sleep measured through a survey | Daily throughout the six week intervention period
  Participants will log their hours of sleep and hours they wear their splint each night to determine if they are able to sleep longer when wearing the splint compared to before they wore the splint. This data will be tracked to ensure the intervention is not decreasing hours of sleep significantly. The change in hours of sleep across the six-week intervention period will be assessed.
Disability of the Arm, Shoulder, and Hand Questionnaire | One time before the intervention begins (During the initial visit)
  Self-administered outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100. This will be used to assess the participant's ability to complete occupation based tasks with their affected hand.
Disability of the Arm, Shoulder, and Hand Questionnaire | One time within a week of completing the six week intervention
  Self-administered outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100. This will be used to assess the participant's ability to complete occupation based tasks with their affected hand.
Number of patients with intact skin integrity of the hands through photographs | Photographs of the hand will be taken one day before the six week intervention begins
  Photographs of the wrist and hand will be taken to assess the skin integrity of the hand that is wearing the splint. Intact skin integrity is indicated by the absence of ulcers, sores, and redness.
Change in the number of patients with intact skin integrity of the hands through photographs | Every other week throughout the intervention period, a total of three times during the intervention which is six weeks long.
  Photographs of the wrist and hand will be taken to assess the skin integrity of the hand that is wearing the splint. Intact skin integrity is indicated by the absence of ulcers, sores, and redness.
Patient satisfaction with splinting process - Individual Interview | Half way through the six week intervention period the participants will be interviewed (at week three)
  The participants will complete a brief 15 minute interview to assess their overall satisfaction with the novel splinting method and splinting intervention. The interview will occur via Zoom or phone call. The participant will answer the following questions:
  1. How do you feel the scanning process went?
  2. Were you uncomfortable at all throughout the scanning process? (ie. Did your arm feel discomfort at any point? If so on a scale from 0-10 what was the discomfort level?)
  3. How do you feel the splint intervention is going?
  4. Do you have any questions or concerns?
Patient satisfaction with splinting process - Individual Interview | Within a week of completing the six week intervention, the participants will be interviewed
  The participants will complete a brief 15 minute interview to assess their overall satisfaction with the novel splinting method and splinting intervention. The interview will occur via Zoom or phone call. The participant will answer the following questions:
  How do you feel the splint intervention went? 2. What would you have wished would have been different throughout this process? 3. Do you feel as though this process was beneficial for you?

CONTACTS AND LOCATIONS:
Locations (1):
- Russell Sage College, Troy, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT05351060/ICF_000.pdf